CLINICAL TRIAL: NCT04482894
Title: Palliative Care Oncology in Patients With Relapsed, Refractory, and High-Risk Leukemias or High-Risk Myelodysplastic Syndrome: Randomized Phase II Study
Brief Title: Palliative Care Oncology in Patients With Relapsed, Refractory, and High-Risk Leukemias or MDS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Karen Ballen, MD, Professor of Medicine, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSR 200133
Record Dates: First submitted 2020-07-08; First posted 2020-07-23 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Leukemia, Acute; AML, Adult; ALL, Adult; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Palliative Care Intervention (Experimental): Participants on this arm will see a palliative care specialist twice a week while they are in the hospital and about every other week when they are out of the hospital. If participants see their oncologist less often than every other week while they're out of the hospital, then visits with the palliative care specialist would be timed to occur on the same day as the oncologist visit. Participants will complete a questionnaire about once a month.
  Interventions: Other: Palliative Care Visits
- Standard Clinical Care (No Intervention): Participants will see a palliative care specialist only if they have a referral from their oncologist according to standard clinical care. Participants on this arm will not be discouraged from requesting a consult.

INTERVENTIONS:
Other: Palliative Care Visits — Regular visits with a palliative (supportive) care specialist
  Arms: Palliative Care Intervention

SUMMARY:
The purpose of this study is to estimate the potential benefit of early and continued palliative care (PC) consultation on end of life issues.

DETAILED DESCRIPTION:
Participants in this study will be randomized to either an intervention group or a standard of care group. Participants in the intervention group will participate in regular visits with a palliative (or supportive) care specialist, while participants in the standard of care group will only see palliative care specialists if the clinician requests a referral. All participants will be asked to complete monthly questionnaires regarding their general well-being.

Participants have a greater chance of being assigned to the intervention group than to the standard of care group. On average, in every 5 people randomized, 3 will be randomized to the intervention and 2 will be randomized to standard of care.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to provide informed consent
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Any of the following:

   1. Patients with a new diagnosis of AML, ALL, high risk myelodysplastic syndrome (MDS), or high risk chronic myelomonocytic leukemia (CMML) who are age 65 and older.

      OR
   2. Patients with relapsed AML, ALL, high risk MDS or high risk CMML, ages 18 and older.

      OR
   3. Patients with refractory AML, ALL, high risk MDS or high risk CMML, ages 18 and older.

Refractory AML/ALL will be defined as persistent leukemia despite two or more cycles of induction chemotherapy.

Refractory MDS will be defined according to the 2006 IWG response criteria Refractory CMML will be based on the assessment of the treating investigator.

Exclusion Criteria:

1. Participants must not have a diagnosis of Acute Promyelocytic Leukemia (APL)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2020-08-19 (Actual); Primary Completion 2025-05-09 (Actual); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Place of death | At the time of death (for participants that die), assessed from enrollment through study completion, an average of 2 years
  Location of death (ICU, inpatient floor, hospice, home)

SECONDARY OUTCOMES:
Overall survival | From enrollment through participant death or end of study from enrollment through participant death or study completion, an average of 2 years.
  Time from enrollment through death (for participants that die)
Duration of hospitalizations | From enrollment through participant death or study completion, an average of 2 years.
  Duration of hospitalizations
Type(s) of hospitalizations | From enrollment through participant death or study completion, an average of 2 years.
  Type(s) of hospitalizations
Frequency of hospitalizations | From enrollment through participant death or study completion, an average of 2 years.
  Frequency of hospitalizations
Emergency department visits | From enrollment through participant death or study completion, an average of 2 years.
  Frequency/Number of emergency department visits
Hospice services use | From enrollment through participant death or study completion, an average of 2 years.
  Dates of use of hospice services
Transfusions | From enrollment through participant death or study completion, an average of 2 years.
  Frequency/number and types of transfusions received
Quality of life measure | At time of enrollment, and then once a month during participation through participant death or study completion, an average of 2 years.
  Quality of life based on FACT-Leukemia questionnaire, scored from 0 to 176, with a higher score indicating better quality of life
Code status change | From enrollment through participant death or study completion, an average of 2 years.
  Dates and types of changes to code status (e.g. Do not rescuscitate (DNR) with details)
Goals of Care (GOC) Discussions | From enrollment through participant death or study completion, an average of 2 years.
  Whether a GOC discussion occurs while on study, and if so, date and location of discussion

CONTACTS AND LOCATIONS:
Overall Officials: Karen Ballen, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No